CLINICAL TRIAL: NCT00377182
Title: A Randomized, Double-blind Study to Evaluate the Safety and Tolerability of the HCV Polymerase Inhibitor Pro-drug in Combination With Pegasys, With or Without Copegus, Versus Pegasys Plus Copegus, in Treatment-naïve Patients With Chronic Hepatitis C, Genotype 1
Brief Title: A Study of Hepatitis C Virus (HCV) Polymerase Inhibitor Pro-Drug in Combination With PEGASYS With or Without COPEGUS in Patients With Chronic Hepatitis C (CHC) Genotype 1 Infection.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PV18369
Record Dates: First submitted 2006-09-15; First posted 2006-09-18 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- PEGASYS with COPEGUS (Active Comparator)
  Interventions: Drug: Copegus; Drug: PEGASYS
- RO5024048 1500mg in combination with PEGASYS (Experimental)
  Interventions: Drug: PEGASYS; Drug: RO5024048 1500mg
- RO5024048 3000mg in combination with PEGASYS (Experimental)
  Interventions: Drug: PEGASYS; Drug: RO5024048 3000mg
- RO5024048 in combination with PEGASYS and COPEGUS (Experimental)
  Interventions: Drug: Copegus; Drug: PEGASYS; Drug: RO5024048 1500mg

INTERVENTIONS:
Drug: Copegus — 1000/1200mg po daily for 4 weeks
  Arms: PEGASYS with COPEGUS; RO5024048 in combination with PEGASYS and COPEGUS
Drug: PEGASYS — 180 micrograms sc weekly for 4 weeks
Drug: RO5024048 1500mg — 1500mg po bid for 4 weeks
  Arms: RO5024048 1500mg in combination with PEGASYS; RO5024048 in combination with PEGASYS and COPEGUS
Drug: RO5024048 3000mg — 3000mg po bid for 4 weeks
  Arms: RO5024048 3000mg in combination with PEGASYS

SUMMARY:
This 4 arm study will compare the safety and tolerability of HCV polymerase inhibitor pro-drug in combination with PEGASYS +/- COPEGUS with the standard of care therapy of PEGASYS + COPEGUS, in treatment-naive patients with CHC, genotype 1. Patients will be randomized to receive 1500mg or 3000mg po bid of HCV polymerase inhibitor pro-drug + PEGASYS, 1500mg of HCV polymerase inhibitor pro-drug + PEGASYS + COPEGUS or PEGASYS + COPEGUS for 4 weeks. All patients who receive at least one dose of study medication will receive open label PEGASYS + Copegus for an additional 44 weeks after the 4 week experimental period. The anticipated time on study treatment is 3-12 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-65 years of age;
* CHC without liver cirrhosis or incomplete/transition to liver cirrhosis, genotype 1;
* chronic liver disease consistent with CHC.

Exclusion Criteria:

* infection with any HCV genotype other than genotype 1;
* previous treatment for CHC;
* medical condition associated with chronic liver disease other than CHC;
* HIV, Hepatitis A, Hepatitis B infection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2006-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) and laboratory parameters. | Week 4, 8 and Week 72

SECONDARY OUTCOMES:
Plasma concentration of HCV polymerase inhibitor | Week 4 and 8
Antiviral activity | Week 4, 8 and Week 72

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- United States (16):
  - La Jolla, California
  - Long Beach, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Aurora, Colorado
  - Bradenton, Florida
  - Gainesville, Florida
  - Chicago, Illinois
  - Novi, Michigan
  - Manhasset, New York
  - New York, New York
  - Chapel Hill, North Carolina
  - Dallas, Texas
  - Fort Sam Houston, Texas
  - Richmond, Virginia
- Santurce, Puerto Rico